CLINICAL TRIAL: NCT00166738
Title: Analysis of Genomic DNA Alterations in Familial Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700834
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; multiple genes; array-comparative genomic hybridization (CGH); genomic DNA; Chinese Han People
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Persons with schizophrenia experience imaginary voices, visions and disorganized thoughts, and are handicapped when it comes to social life, which is detrimental to the affected individuals and the community. Although the pathogenesis of this mental disease has not been clearly elucidated, much evidence suggests that inheritance is of major etiological importance and multiple genetic components are implicated. Previous linkage studies of familial schizophrenia have led to the successful identification of numerous susceptibility loci covering many of the human chromosomes, including chromosome 1q, 5q, 6p22, 6p24, 8q21, 13q32, 15q13-14 and 22q11, etc. Necessities for further identification of candidate genes involved in familial schizophrenia by taking a genome-wide approach are listed as follows:

1. given that multiple genes are responsible for this disease, it is of critical interest to view the complete molecular profiling of schizophrenia's genome;
2. identification of promising schizophrenia candidate genes by genome-wide scanning will facilitate the development of molecular markers and provide a more objective and effective assessment method in psychotic diagnosis and prognosis;
3. prevention of the onset of this disorder will be improved by early classification of individuals bearing strong genetic loading for schizophrenia as a high risk population;
4. making a breakthrough into the investigation of schizophrenia pathogenesis by the characterization of susceptible genes found by genome-wide exploring.

Array-based comparative genomic hybridization (CGH) allows high-throughput genome-wide survey for DNA copy number aberrations, providing a powerful tool for investigating genetic disorders and for developing diagnostic and therapeutic targets. Arrays used in this study consist of approximately 43,000 60-mer oligonucleotide probes that span coding and noncoding regions of the whole human genome with an average spatial resolution of around 35 kb. Furthermore, the sensitivity of these arrays is capable of detecting and mapping regions of single-copy losses, homozygous deletions, and amplicons of various sizes even when using full-complexity genomic samples. In this study, the investigators will conduct an array-based comparative genomic hybridization (CGH) with genomic DNA of many affected members from "schizophrenia families" (the investigators classified families according to the presence or absence of two or more affected members) to identify a set of candidate genes associated with this disease. It is hoped that the results obtained from this study will improve the accuracy and efficiency of psychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Familial schizophrenia
* Over 9 years of education

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University
Locations (1):
- Hai-Gwo Hwu, Taipei, Taiwan